CLINICAL TRIAL: NCT04700241
Title: Acute Effects of Inorganic Nitrate on Brain Insulin-sensitivity in Abdominally Obese Men
Brief Title: Nitrate and Brain Insulin-Sensitivity
Acronym: NO-BRAINS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: METC 20-0.78
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-04

CONDITIONS: Nitrate; Brain Insulin-sensitivity; Vascular Function
MeSH Terms: interventions — potassium nitrate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potassium nitrate (Active Comparator): During this experimental day, men will receive 10 mmol of potassium nitrate
  Interventions: Dietary Supplement: Potassium nitrate
- Placebo (Placebo Comparator): During this experimental day, men will receive an isomolar dose of potassium chloride
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Potassium nitrate — Acute intervention (5.5 hours)
  Arms: Potassium nitrate
Dietary Supplement: Placebo — Acute intervention (5.5 hours)
  Arms: Placebo

SUMMARY:
Disturbances in brain insulin-sensitivity are not only observed in abdominal obesity and type 2 diabetes mellitus (T2D), but also during brain aging and in dementia. Inorganic nitrate may improve brain insulin-sensitivity, which can be quantified by measuring the gray-matter cerebral blood flow (CBF) response to intranasally administered insulin, through beneficial effects on brain vascular function. Therefore, we now hypothesize that inorganic nitrate, which can be found in several vegetables such as beetroot, improves brain insulin-sensitivity, as assessed by the gray-matter CBF response to intranasally administered insulin, in abdominally obese men.

ELIGIBILITY:
Inclusion Criteria:

* Men;
* Aged between 18 - 60 years;
* Waist circumference > 102 cm (abdominally obese);
* Fasting plasma glucose ≤ 7.0 mmol/L;
* Fasting serum total cholesterol ≤ 8.0 mmol/L;
* Systolic blood pressure < 160 mmHg and diastolic blood pressure < 100 mmHg;
* Stable body weight (weight gain or loss < 3 kg in the past three months);
* Willingness to give up being a blood donor from 8 weeks before the start of the study, during the study and for 4 weeks after completion of the study;
* Willingness not to use antibacterial mouth wash or toothpaste, chewing-gum and tongue-scraping a week before the study;
* No difficult venipuncture as evidenced during the screening visit.

Exclusion Criteria:

* Women;
* Left-handedness;
* Current smoker, or smoking cessation < 12 months;
* Diabetic patients;
* Familial hypercholesterolemia;
* Abuse of drugs;
* More than 3 alcoholic consumptions per day;
* Use of products or dietary supplements known to interfere with the main outcomes as judged by the principal investigators;
* Use medication to treat blood pressure, lipid or glucose metabolism;
* Pharmacological treatment advised based on the Dutch general practitioners' association (NHG) for cardiovascular risk management;
* Use of an investigational product within another biomedical intervention trial within the previous 1-month;
* Severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases and rheumatoid arthritis;
* Active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebrovascular accident;
* Specific contra-indications for MRI imaging, including pacemakers, surgical clips/material in body, metal splinters in eye, claustrophobia, or tattoos in the facial area, such as permanent make-up.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Brain insulin sensitivity | Change from placebo intervention at 2 hours after supplement intake
  MRI arterial spin labeling, cerebral blood flow measurements before and after a nasal insulin spray

SECONDARY OUTCOMES:
Brain vascular function | Change from placebo intervention at 2 hours after supplement intake
  MRI arterial spin labeling, cerebral blood flow measurements
Vascular function markers | Change from fasting at 4 hours after supplement intake
  Flow-mediated vasodilation (FMD) of the brachial and femoral artery
Cold pressure test | Change from placebo at 4 hours after supplement intake
  Carotid artery response to cold pressure test
Cardiometabolic risk markers (1) | Change from placebo at 4 hours after supplement intake
  Plasma markers for low-grade systemic inflammation (CRP)
Cardiometabolic risk markers (2) | Change from placebo at 4 hours after supplement intake
  Plasma marker for endothelial dysfunction (NOx)
Cardiometabolic risk markers (3) | Change from placebo at 4 hours after supplement intake
  Office blood pressure
Cardiometabolic risk markers (4) | During the 5.5 hours following supplement intake
  Plasma brain derived neurotrophic factor (BDNF)
Postprandial metabolism (1) | During the 5.5 hours following supplement intake
  Serum lipid metabolism
Postprandial metabolism (2) | During the 5.5 hours following supplement intake
  Plasma glucose metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Joris, Dr, Principal Investigator — Maastricht University; Ronald P.M. Mensink, Dr, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kleinloog JPD, Mensink RP, Smeets ETHC, Ivanov D, Joris PJ. Acute inorganic nitrate intake increases regional insulin action in the brain: Results of a double-blind, randomized, controlled cross-over trial with abdominally obese men. Neuroimage Clin. 2022;35:103115. doi: 10.1016/j.nicl.2022.103115. Epub 2022 Jul 14. PMID 35843050